CLINICAL TRIAL: NCT06340100
Title: Association of History of Concussion With Vestibular Impairment and Cognitive Function in Sports Athletes
Status: Recruiting | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/MS-PT/01832
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Concussion, Mild; Vestibular Impairment; Cognitive Impairment
MeSH Terms: conditions — Brain Concussion; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- concussed contact sports athlete: Informed Consent: Participants are provided with information about the study, including its purpose, procedures, potential risks, and benefits. They are given the opportunity to ask questions and provide informed consent before participating.
  Baseline Assessments: Before any interventions or assessments, participants undergo baseline evaluations of their vestibular function and cognitive abilities. This helps establish a starting point for comparison and allows researchers to identify any pre-existing impairments.
  Concussion History Questionnaires: Participants complete questionnaires or interviews to provide detailed information about their history of concussions, including the number, severity, and timing of each injury.
  Interventions: Other: find association between vestibular impairment , cognitive fiunction with concussin

INTERVENTIONS:
Other: find association between vestibular impairment , cognitive fiunction with concussin — SCOAT 6 is a standardized tool used for evaluating athletes suspected of having a concussion. It includes a variety of components such as symptom evaluation, cognitive assessment, balance evaluation, and a neck examination. it helps in assessing the severity of the injury, tracking recovery, and making return-to-play decisions. Dr. Robert Cantu, a prominent figure in sports concussion research, has proposed guidelines for the management of concussions. These guidelines typically involve recommendations for the evaluation, treatment, and return-to-play decisions for athletes who have sustained concussions
  Other Names: identify concussion and find asociation through scoat 6 ad Cantu

SUMMARY:
This study investigates the potential relationship between prior concussions and their impact on both vestibular function and cognitive abilities in athletes participating in sports.

DETAILED DESCRIPTION:
The association of a history of concussions with vestibular impairment and cognitive function in sports athletes is a significant area of research due to the potential long-term consequences of head injuries in contact sports.

Vestibular impairment refers to disruptions in the balance and spatial orientation system of the inner ear, which can result from head trauma. Cognitive function encompasses various mental processes, including memory, attention, and decision-making, which may be affected by concussions.

This study aims to examine how prior concussions relate to both vestibular impairment and cognitive function in athletes participating in sports. Researchers typically employ a combination of self-reported concussion history, clinical assessments of vestibular function, and standardized cognitive tests to evaluate participants.

Findings from such studies can provide valuable insights into the potential effects of concussions on athletes' balance, spatial awareness, and cognitive abilities. Understanding these associations can inform concussion management protocols, rehabilitation strategies, and preventive measures in sports settings.

Furthermore, this research may contribute to the development of targeted interventions aimed at improving vestibular rehabilitation and cognitive training for athletes with a history of concussions. By identifying and addressing these potential deficits early, athletes may reduce their risk of long-term complications and optimize their performance and well-being in sports.

ELIGIBILITY:
Inclusion Criteria:

* athletes actively involved in sports at age of 18 to 35
* active players in contact sports

Exclusion Criteria:

* Concussion other than sports
* History of recent fractures.
* Participants having neurological deficits

Ages: 18 Years to 36 Years | Sex: All
Age Groups: Adult
Study Population: This includes information such as age, gender, and ethnicity of the athletes. Understanding the demographics of the population helps in assessing the generalizability of the study findings across different groups.
  The number, severity, and timing of previous concussions experienced by each athlete. This helps in stratifying the participants based on concussion history and assessing potential cumulative effects.
  Pre-existing medical conditions, history of previous injuries (e.g., musculoskeletal injuries), and baseline cognitive and physical performance measures. This information allows for controlling potential confounding variables and assessing the impact of concussion independently.
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2024-03-23 (Actual); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
CANTU | 3 DAYS
  The Cantu guidelines, named after Dr. Robert Cantu, are a set of recommendations for the management of concussions in sports. Dr. Cantu, a renowned neurosurgeon and concussion expert, has contributed significantly to the understanding and treatment of concussions, particularly in the field of sports medicine. While there isn't a single document titled "Cantu Description," Dr. Cantu's work encompasses various aspects of concussion management, including diagnosis, treatment, and return-to-play protocols.
Sports concussion office assesment tool 6 | 3-30days
  SCOAT 6 is a standardized tool used for evaluating athletes suspected of having a concussion. It includes a variety of components such as symptom evaluation, cognitive assessment, balance evaluation, and a neck examination. it helps in assessing the severity of the injury, tracking recovery, and making return-to-play decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Maheen gul, MSSPT*, Principal Investigator — Riphah International University
Locations (1):
- HAYATABAD Sports complex, Peshawar, Khyber Pakhtun Khawan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitney SL, Eagle SR, Marchetti G, Mucha A, Collins MW, Kontos AP; CARE Consortium Investigators. Association of acute vestibular/ocular motor screening scores to prolonged recovery in collegiate athletes following sport-related concussion. Brain Inj. 2020 May 11;34(6):840-845. doi: 10.1080/02699052.2020.1755055. Epub 2020 Apr 21. PMID 32315218
- [Background] Taylor KM, Kioumourtzoglou MA, Clover J, Coull BA, Dennerlein JT, Bellinger DC, Weisskopf MG. Concussion History and Cognitive Function in a Large Cohort of Adolescent Athletes. Am J Sports Med. 2018 Nov;46(13):3262-3270. doi: 10.1177/0363546518798801. Epub 2018 Sep 19. PMID 30230912
- [Background] Price AM, Knell G, Caze TJ 2nd, Abt JP, Loveland D, Burkhart SO. Exploring Vestibular/Ocular and Cognitive Dysfunction as Prognostic Factors for Protracted Recovery in Sports-Related Concussion Patients Aged 8 to 12 Years. Clin J Sport Med. 2022 Jul 1;32(4):408-414. doi: 10.1097/JSM.0000000000000975. Epub 2021 Sep 8. PMID 34516435
- [Background] Yorke AM, Smith L, Babcock M, Alsalaheen B. Validity and Reliability of the Vestibular/Ocular Motor Screening and Associations With Common Concussion Screening Tools. Sports Health. 2017 Mar/Apr;9(2):174-180. doi: 10.1177/1941738116678411. Epub 2016 Nov 11. PMID 27834667
- [Background] Eagle SR, Nindl BC, Johnson CD, Kontos AP, Connaboy C. Does Concussion Affect Perception-Action Coupling Behavior? Action Boundary Perception as a Biomarker for Concussion. Clin J Sport Med. 2021 May 1;31(3):273-280. doi: 10.1097/JSM.0000000000000731. PMID 30829684
- [Background] Zhang Y, Ma Y, Chen S, Liu X, Kang HJ, Nelson S, Bell S. Long-Term Cognitive Performance of Retired Athletes with Sport-Related Concussion: A Systematic Review and Meta-Analysis. Brain Sci. 2019 Aug 13;9(8):199. doi: 10.3390/brainsci9080199. PMID 31412586
- [Background] Louey AG, Cromer JA, Schembri AJ, Darby DG, Maruff P, Makdissi M, Mccrory P. Detecting cognitive impairment after concussion: sensitivity of change from baseline and normative data methods using the CogSport/Axon cognitive test battery. Arch Clin Neuropsychol. 2014 Aug;29(5):432-41. doi: 10.1093/arclin/acu020. Epub 2014 May 9. PMID 24813184
- [Background] Harmon KG, Clugston JR, Dec K, Hainline B, Herring S, Kane SF, Kontos AP, Leddy JJ, McCrea M, Poddar SK, Putukian M, Wilson JC, Roberts WO. American Medical Society for Sports Medicine position statement on concussion in sport. Br J Sports Med. 2019 Feb;53(4):213-225. doi: 10.1136/bjsports-2018-100338. PMID 30705232
- [Background] Bryan MA, Rowhani-Rahbar A, Comstock RD, Rivara F; Seattle Sports Concussion Research Collaborative. Sports- and Recreation-Related Concussions in US Youth. Pediatrics. 2016 Jul;138(1):e20154635. doi: 10.1542/peds.2015-4635. Epub 2016 Jun 20. PMID 27325635
- [Background] Kerr ZY, Roos KG, Djoko A, Dalton SL, Broglio SP, Marshall SW, Dompier TP. Epidemiologic Measures for Quantifying the Incidence of Concussion in National Collegiate Athletic Association Sports. J Athl Train. 2017 Mar;52(3):167-174. doi: 10.4085/1062-6050-51.6.05. Epub 2016 Jun 22. PMID 27331336